CLINICAL TRIAL: NCT05022511
Title: Three Birds With One Stone: a Randomised Intervention Study to Increase Participation in Cervical and Colorectal Cancer Screening Among Women Attending Breast Cancer Screening
Brief Title: Three Birds With One Stone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Three birds with one stone
Record Dates: First submitted 2021-08-10; First posted 2021-08-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-09

CONDITIONS: Uterine Cervical Cancer; Uterine Cervix Cancer; Uterine Cervical Neoplasm; Colorectal Neoplasms; Colorectal Cancer; Colorectal Carcinoma; Mass Screening; Early Detection of Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): All women aged 50-69 years attending breast cancer screening in the intervention unit on an intervention day. They will all be offered to receive information on their screening status in cervical cancer og colorectal cancer screening.
  Women aged 50-64 years, who have not had a cervical cytology sample taken within 5 years and 6 months will be offered to receive a self-sample device for high risk human papilloma virus (hrHPV) screening by mail, or reminded to see her general practitioner (GP) to have a conventional cervical cytology sample taken.
  Women aged 50-69 years, who have not had a Faecal Immunochemical Test (FIT) within 2 years and 4.5 months will be offered to receive a new self-sampling kit for FIT.
  Interventions: Behavioral: Screening status
- Control group (No Intervention): Women in the control group will receive standard screening offers according to the national screening programme.

INTERVENTIONS:
Behavioral: Screening status — Women are offered check-up on screening status in both CCU and CRC screening. If a woman is not up to date in one or both screening programmes, she will be offered a self-sampling device and/or a FIT kit.
  Arms: Intervention group

SUMMARY:
The overall aim of the study is to increase participation rates in cervical cancer (CCU) and colorectal cancer (CRC) screening programmes in Denmark by offering home-based CCU and CRC screening to women who are overdue for one or both screening programmes when attending breast cancer screening

DETAILED DESCRIPTION:
A cluster-randomised public health trial will take place in Central Denmark Region (CDR) targeting women attending breast cancer screening. Five breast cancer screening units serve women five days a week, and all five units will be included in the study and randomly allocated to an equal amount of intervention days. On the intervention days, the other four units will serve as the control group, providing a randomisation ratio of 1:4.

On the intervention days, a research assistant will ask the women aged 50-69 years if they are interested in having a check up on their screening status with CCU and CRC screening. If the woman has not participated timely, she will be offered to receive a test-kit corresponding to CRC screening and/or to receive a self-sample device for CCU screening (or reminded to call her general practitioner (GP) to have a conventional cervical cytology sample taken).

If the woman accepts a self-sample kit for CCU and/or CRC screening, she will receive it by mail together with written instructions, picturebased user instructions, information on national recommendation for cancer screening and a pre-paid, pre-addressed envelope for returning the sample to the laboratory.

The result of the test will be sent to the women by digital mail as well as passed on to her GP.

Clinical management in case of a positive test result will follow national guidelines corresponding to CCU and CRC screening programmes.

Women in the control group will receive standard screening offers according to the national screening programmes.

All women entering a breast cancer screening unit in CDR on a intervention day (intervention + control units) will be sent a survey asking their experience with breast cancer screening a few days after breast cancer screening. The women in the intervention group will be asked about the acceptability of the intervention as well.

27500 women must be included, of which 5500 women will be in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

Women aged 50-69 years attending breast cancer screening in Central Denmark Region on selected days.

* In CCU screening: women aged 50-64 years will be classified as overdue if they have not had a cervical sample within the last 5 years and 6 months
* In CRC screening: women aged 50-69 years will be classified as overdue, if they have not had a FIT within the last 2 years and 4.5 months despite an invitation.

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27099 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Coverage | 180 days after participating in breast cancer screening
  Difference in overall coverage og CCU/CRC screening six months after the intervention between control and intervention group
Participation | 180 days after participating in breast cancer screening
  Difference between intervention and control group in proportion of women participating in CCU and CRC screening after 180 days for those overdue with CCU/CRC screening at the intervention

SECONDARY OUTCOMES:
Prevalence of hrHPV in self-samples in CCU screening | After study completion, expected to be 1 year
Rate of compliance to follow-up in CCU screening | Within 180 days after a positive hrHPV self-sample
  A GP collected sample after a hrHPV positive self-sample
Register-based screening history of self-samplers in CCU screening | After test completion. expected to be 1 year
  "Under-screened" defined as screened at least once with in the last 10 years prior to the intervention. "Un-screened" defined as no screening sample with in the last 10 years prior to the intervention.
Prevalence of colposcopies after CCU screening | Within 180 days after a positive hrHPV self-sample
Incidence of CIN2+ | Within 180 days after a positive hrHPV self-sample
Incidence of hrHPV positive cases in women 60-64 years after 12 months with an initial negative hrHPV sample in CCU screening | After test completion, expected to be 1 year
Prevalence of positive FIT cases after CRC screening for those overdue at the intervention date | After test completion, expected to be 1 year
Histology (number of adenomas, cancer) after a positive FIT in CRC screening | After test completion, expected to be 1 year
Register-based screening history in CRC screening | After test completion, expected to be 1 year
  "Under-screened" defined as at least one FIT, but none with the last 2 years and 4.5 months. "Un-screened" defined as no previous FIT despite invitation
Rate of compliance to follow-up with colonoscopy after a positive FIT | Within 60 days from a positive FIT

OTHER OUTCOMES:
Proportion of women accepting a check up on CCU and CRC screening status | At end of enrollment
  Process outcome within the intervention group
Proportion of women overdue with CCU and/or CRC screening | At end of enrollment
  Process outcome within the intervention group
Proportion of women accepting a test-kit | At end of enrollment
  Process outcome within the intervention group
Proportion of women not returning a test kit | At end of enrollment
  Process outcome within the intervention group
Previous screening history, previous cancer diagnoses, socioeconomic data (age, ethnicity, marital status, educational status) and inflammatory bowel disease | At end of enrollment
  To test if the randomisation succeeded
Survey evaluation | At end of enrollment
  Evaluation regarding the acceptability of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Berit Andersen, Prof., MD, Head of Department, Study Chair — Department of Public Health Programmes and University Clinic for Cancer Screening, Randers Regional Hospital and Department of Clinical Medicine, Aarhus University
Locations (1):
- Anne Dorte Lerche Helgestad, Randers, Denmark

REFERENCES:
- [Derived] Helgestad ADL, Larsen MB, Njor S, Tranberg M, Petersen LK, Andersen B. Increasing coverage in cervical and colorectal cancer screening by leveraging attendance at breast cancer screening: A cluster-randomised, crossover trial. PLoS Med. 2024 Aug 13;21(8):e1004431. doi: 10.1371/journal.pmed.1004431. eCollection 2024 Aug. PMID 39137185
- [Derived] Helgestad ADL, Larsen MB, Njor S, Tranberg M, Petersen LK, Andersen B. Three birds with one stone: a protocol for a randomised intervention study to increase participation in cervical and colorectal cancer screening among women attending breast cancer screening. BMJ Open. 2022 Sep 22;12(9):e062824. doi: 10.1136/bmjopen-2022-062824. PMID 36137619